CLINICAL TRIAL: NCT04385043
Title: Efficacy and Safety of Hyperimmune Plasma Treatment in Patients With COVID-19 Severe Infection
Brief Title: Hyperimmune Plasma in Patients With COVID-19 Severe Infection
Acronym: COV2-CP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Collaborators: Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other); Azienda Sanitaria Provinciale Di Catanzaro (Other); Annunziata Hospital, Cosenza, Italy (Other); Azienda Ospedaliera Bianchi-Melacrino-Morelli (Other)
Responsible Party: Principal Investigator, Luca Gallelli, MD, University of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Covid-19 convalescent plasma
Record Dates: First submitted 2020-05-04; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: severe Covid-19; severe coronavirus-2; plasma hyperimmune; convalescent plasma
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plasma-hyperimmune (Experimental): enrolled patients (n=200) with severe Covid-19 infection will receive a treatment with plasma hyperimmune add on to the standard therapy
  Interventions: Other: plasma hyperimmune; Drug: standard therapy
- standard therapy (Active Comparator): enrolled patients (n=200) with severe Covid-19 infection will receive a treatment with the standard therapy
  Interventions: Drug: standard therapy

INTERVENTIONS:
Other: plasma hyperimmune — patients will receive this as add on therapy
  Arms: plasma-hyperimmune
Drug: standard therapy — patients will receive only standard therapy for Covid-19 infection

SUMMARY:
Passive immunotherapy through plasma infusion of convalescent subjects - convalescent plasma - or "hyperimmune" plasma was one of the most widespread and effective anti-infective treatments in the pre-antibiotic era and one of the founding pillars of immunology, and has also been used during the SARS (2002-2003) and Ebola (2014-2016) viral epidemy for which there were no alternative immunoprophylactic or therapeutic interventions.

To date, there are not proven etiological therapies for SARS-CoV-2 infection, the agent responsible for the disease called Covid-19. Among those subjected to clinical studies during the current epidemic in China, hyperimmune plasma appears to be one of the most rational and promising.

The objective of this study will be to evaluate the efficacy and safety of the hyperimmune plasma administered add-on to the anti-Covid-19 treatment (standard therapy) according to clinical practice in patients with severe Covid-19 infection, compared to patients with severe Covid-19 infection treated only with standard therapy.

DETAILED DESCRIPTION:
Passive immunotherapy through plasma infusion of convalescent subjects - convalescent plasma - or "hyperimmune" plasma was one of the most widespread and effective anti-infective treatments in the pre-antibiotic era and one of the founding pillars of immunology. Immunoprophylaxis represents an irreplaceable protection for post-exposure prevention of several viral infections such as measles, hepatitis B and rabies. Recently, the use of convalescent plasma for therapeutic purposes has been re-evaluated during the SARS (2002-2003) and Ebola (2014-2016) epidemic caused by serious viral infections for which there were no immunoprophylactic or therapeutic interventions. alternative. The results of these experimental interventions, despite the limited number and the often anecdotal character, have shown promise even if not conclusive. In the case of SARS, the first human respiratory disease caused by a Coronavirus, treatment with convalescent plasma was associated with a 23% reduction in mortality and with the best results if administered at an early stage of the disease. In addition, all the evidence available in the literature has confirmed the safety of convalescent plasma treatments, in line with what has already been observed in the transfusion practice with Fresh Frozen Plasma.

As is known, there are currently no proven etiological therapies to combat SARS-CoV-2 infection, the agent responsible for the disease called Covid-19. Among those subjected to clinical studies during the current epidemic in China, hyperimmune plasma appears to be one of the most rational and promising.

Waiting for the numerous clinical trials underway especially in Asia and accessible on the website http://apps.who.int/trialsearch/default.aspx to define if and to what extent this therapeutic contribution improves the prognosis of patients suffering from serious forms of infections from SARS-Co-2, the clinical guidelines of the People's Republic of China, already provide for the use of hyperimmune plasma with the indication "in rapidly progressive disease, severe and very severe form" and by the FDA .

As regards the technical protocols for the preparation of hyperimmune plasma for clinical use in the literature, precise references are available in particular for the preparation, qualification, viral inactivation and dosage of hyperimmune plasma for the treatment of viral epidemic infections such as MERS and Ebola and which can also be validated and used for the preparation of plasma from convalescent patients for Covid-19.

From the above, the objective of this study will be to evaluate the efficacy and safety of the hyperimmune plasma administered add-on to the anti-Covid-19 treatment (standard therapy) according to clinical practice in patients with severe Covid-19 infection, compared to patients with severe Covid-19 infection treated only with standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* inclusion criteria for donors: null-gravid, with a negative history of transfusion of blood components; possibility to sign the informed consent
* inclusion criteria for Covid-19 infected patients: serious Covid-19 infection, possibility to sign the informed consent (also through the legal tutor)

Exclusion Criteria:

* exclusion criteria for donors: presence of pregnancy, recent history of transfusion of blood components, < 18 years.
* exclusion criteria for Covid-19 infected patients: non serious Covid-19 infection, impossibility to sign the informed consent (also through the legal tutor)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
decrease in mortality | 30 days
  Statistically significant reduction (P <0.05) of mortality in the group of patients treated with hyperimmune plasma vs patients treated with standard therapy.

SECONDARY OUTCOMES:
lymphocytes | 7 and 14 days
  Statistically significant increase (P <0.05) of lymphocyte levels after 7 and 14 days after the start of treatment with hyperimmune plasma (treated group), compared to the control group.
PCR levels vs control | 7 and 14 days
  Statistically significant reduction (P <0.05) of plasma levels of reactive protein C (expressed as mg/L), 7 and 14 days after the start of treatment with hyperimmune plasma vs standard therapy (group control)
PCR levels vs before treatment | 7 and 14 days
  Statistically significant reduction (P <0.05) of plasma levels of reactive protein C (expressed as mg/L), 7 and 14 days after the start of treatment with hyperimmune plasma vs the same patients before the beginning of the treatment
AB levels and clinical improvement | 30 days
  Significant Correlation (P<0.05) between hyperimmune plasma antibody levels and clinical improvement time (expressed in days)
Inflammatory cytokines vs controls | 7 and 14 days
  Statistically significant reduction (P <0.05) of plasma levels of IL-6 (expressed as pg/mL) and TNF-alpha (expressed as pg/mL), 7 and 14 days after the start of treatment with hyperimmune plasma vs standard therapy (group control)
Inflammatory cytokines vs before treatment | 7 and 14 days
  Statistically significant reduction (P <0.05) of plasma levels of IL-6 (expressed as pg/mL) and TNF-alpha (expressed as pg/mL), 7 and 14 days after the start of treatment with hyperimmune plasma vs the same patients before the beginning of the treatment

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Azienda Ospedaliera Policlinico Mater Domini, Catanzaro
  - Azienda Ospedaliera Pugliese Ciaccio Catanzaro, Catanzaro
  - Azienda Ospedaliera Annunziata, Cosenza
  - Azienda Sanitaria Provinciale, Crotone
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Azienda Sanitaria Provinciale, Vibo Valentia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marano G, Vaglio S, Pupella S, Facco G, Catalano L, Liumbruno GM, Grazzini G. Convalescent plasma: new evidence for an old therapeutic tool? Blood Transfus. 2016 Mar;14(2):152-7. doi: 10.2450/2015.0131-15. Epub 2015 Nov 6. PMID 26674811
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Result] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Result] Linee Guida Cinesi sulla Gestione di COVID-19 Versione 7° Pubblicate in data 3/3/2020 dalla Commissione della Salute Nazionale della R.P.C..
- [Result] Arabi Y, Balkhy H, Hajeer AH, Bouchama A, Hayden FG, Al-Omari A, Al-Hameed FM, Taha Y, Shindo N, Whitehead J, Merson L, AlJohani S, Al-Khairy K, Carson G, Luke TC, Hensley L, Al-Dawood A, Al-Qahtani S, Modjarrad K, Sadat M, Rohde G, Leport C, Fowler R. Feasibility, safety, clinical, and laboratory effects of convalescent plasma therapy for patients with Middle East respiratory syndrome coronavirus infection: a study protocol. Springerplus. 2015 Nov 19;4:709. doi: 10.1186/s40064-015-1490-9. eCollection 2015. PMID 26618098
- [Result] Dean CL, Hooper JW, Dye JM, Zak SE, Koepsell SA, Corash L, Benjamin RJ, Kwilas S, Bonds S, Winkler AM, Kraft CS. Characterization of Ebola convalescent plasma donor immune response and psoralen treated plasma in the United States. Transfusion. 2020 May;60(5):1024-1031. doi: 10.1111/trf.15739. Epub 2020 Mar 4. PMID 32129478